CLINICAL TRIAL: NCT01474447
Title: The Research Protocol: The Effect of Grinberg Method (GM) Intervention on Low-back Pain (LBP) and Improving the Quality of Life
Brief Title: The Effect of Grinberg Method (GM) Intervention on Low-back Pain (LBP) and Improving the Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-11-SB-541-CTIL
Record Dates: First submitted 2011-11-02; First posted 2011-11-18 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Low Back Pain (LBP)
Keywords: low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Grinberg Method (Experimental)
  Interventions: Behavioral: Grinberg Method

INTERVENTIONS:
Behavioral: Grinberg Method — The GM is a methodology of attention that teaches through expanding and focusing body attention to create a change and an improvement in pain and in quality of life. The method focuses on the way in which we experience pain, and offers an approach that trains people to use their attention and will in order to turn an unwanted experience that causes suffering, into a controlled experience in which they can take responsibility on the way they react to an existing pain. The method uses attention in order to learn the fixed ways in which we respond to pain in our body: where we focus our attention, what is the level of tension in our muscles, how we breathe and relax and more. It gives simple and effective tools to control all these, in order to create optimal conditions in the body to utilize its natural potential to recover and recuperate

SUMMARY:
The purpose of the research is to check the efficiency of practicing the tools of the Grinberg method (GM) in reducing Low-back Pain (LBP), reducing limitations in movement as a result of the pain, and improving the general quality of life.

The hypothesis suggests that by learning to perceive pain differently, the level of pain will reduce and general well-being improved.

DETAILED DESCRIPTION:
The research will include 140 patients, who attended the pain clinic due to chronic LBP. Any change in the pharmacological regimen will be done with consult of the tending doctor and the change will be reported.

Tools and Methods A patient, whom volunteers to take part in the research, will be invited to the Ichilov Pain clinic in order to fill-in questionnaires and sign an informed consent form.

Each participant in the experiment group will participate in a series of 6 sessions lasting 1 hour each, extending between 6 to 8 consecutive weeks, with one of the qualified GM practitioners partaking in the experiment. Each participant will have all their sessions with the same GM practitioner throughout the experiment. Immediately after the last session, the participants will fill-in the same questionnaires given at the beginning of the experiment. The non-GM intervention group will answer the questionnaires after 6-8 weeks of pharmacological treatment only.

Questionnaires:

* General Details and Pain Questionnaire
* SF-MPQ Short Form McGill Pain Questionnaire, Ronald Melzack
* RMDQ - Roland Morris Disability Questionnaire
* SF 36 - The Short Form Health Survey

ELIGIBILITY:
Inclusion Criteria:

* Women and men, age range 18-65; patients of the Ichilov Pain clinic, who suffer from chronic LBP that lasts over 3 months and that appears several times a week.
* LBP which is localized between the 12th rib and the inferior gluteal folds, with or without leg pain. The LBP may be non-specific, mechanical or radicular.

Exclusion Criteria:

* Patients with malignancy and/or other life threatening conditions
* Diabetic patients
* Patients with fibromyalgia
* Pregnancy
* Paralysis
* Patients with obesity
* Patients that underwent organ transplantation
* Severe osteoporosis
* Patients that are scheduled to receive spinal cord injections during the research
* Patients that received less than 4 weeks before the research, other pain interventions than the standard of care treatment such as: alternative medicine (acupuncture, shiatsu, massage, reflexology, homeopathy etc'); physiotherapy, chiropractic, hydrotherapy, bio-feedback, osteopathy and others.
* Patients with severe mental disorders (such as schizophrenia, bipolar disorder, suicidal tendencies etc')
* Pain lasting less than 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
pain questionnaires that will assess the improvement on back pain in patients treated with the Grinberg method | change of pain from baseline and after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Silviu Brill, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Pain Medicine Unit, Tel Aviv, Israel